CLINICAL TRIAL: NCT05152173
Title: Phase 2, Double-blind, Randomized, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of EN3835 vs Placebo in the Treatment of Plantar Fibromatosis
Brief Title: Efficacy, Safety, and Tolerability, of EN3835 vs Placebo in the Treatment of Plantar Fibromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3835-222
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fibromatosis
MeSH Terms: conditions — Fibromatosis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EN3835 Group (Experimental): Participant will receive a maximum dose of up to 1.8mg of EN3835 injection
  Interventions: Biological: EN3835
- Placebo Group (Placebo Comparator): Participant will receive a maximum dose of up to 1.8mg of Placebo injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: EN3835 — Participant will receive a maximum dose of up to1.8mg of EN3835 injection
  Arms: EN3835 Group
Other: Placebo — Participant will receive a maximum dose of up to1.8mg of Placebo injection
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of up to 2 treatments of EN3835 vs placebo in participants with plantar fibromatosis.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of plantar fibromatosis AND have at least 1 measurable, hard or firm, palpable fibrous nodule on clinical examination.
2. Has no significant medical history or examination findings related to the participant's plantar nodule(s), which in the investigator's opinion, would make the participant unsuitable for study intervention administration.
3. Agree not to use opioids during the study period and has not used opioids 2 weeks before the Screening Visit.
4. Agree to not initiate or change use of orthotics or inserts designed to relieve symptoms of plantar fibromatosis during the study period.
5. If female, be of non-childbearing potential (history of hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal with no history of menstrual flow in the 12 months prior to the Screening Visit); or, if of childbearing potential, be non-pregnant, non-lactating and agree to use effective contraception when with a male partner for the duration of the study and for 28 days after any active treatment period.
6. Willing and able to comply with all protocol required visits and assessments.
7. Be adequately informed and understand the nature and risks of the study and be able to provide consent.

Exclusion Criteria:

1. Has the presence of non-plantar fibromatosis-related nodules on the foot/feet (eg, neurofibroma, rhabdomyosarcoma, liposarcoma, neurilemmomas, rheumatoid nodules, desmoid tumors, or malignant soft tissue lesions of the foot or ankle).
2. Has any musculoskeletal, neuromuscular, neurosensory, other neurological or related disorder that affects the participant's use of his or her feet and/or would impair his/her completion of study assessments as determined by the investigator.
3. Has a known allergy to collagenase or any other excipient of EN3835.
4. Has a known coagulation disorder or is taking any medications that would increase the risk of bleeding (except <150mg of aspirin daily), 7 days prior to first injection and for the duration of the study.
5. Has concurrent diseases that might interfere with the conduct of the study, confound the interpretation of the study results or endanger the participant's well-being. If there is a history of such disease and the condition has been stable for greater than one year and is judged by the investigator not to interfere, the participant may be included, with the documented approval of the Medical Monitor.
6. Is from a vulnerable population, as defined by the US Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full-time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the IRB/IEC.
7. Has any other condition(s) that, in the investigator's opinion, might indicate the participants to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Mean Change between EN3835 and placebo in the Foot Function Index (FFI) pain subscale | Baseline (Day1) to Day 57
  Mean change on the foot pain subscale (total score on 9 items) of the FFI ranging from 0 ("None") to 4 ("Extreme").

SECONDARY OUTCOMES:
Mean Change with EN3835 and placebo in the FFI pain subscale | Mean Change from Baseline (Day 1) to Days 15, 29, 43, and 57
  Mean change on the foot pain subscale (total score on 9 items) of the FFI ranging from 0 ("None") to 4 ("Extreme").
Mean change between EN3835 and placebo on the total score of the FFI pain and difficult subscales (combined) | Baseline (Day 1) to Day 57
  Mean change between EN3835 and placebo on the total score of the FFI pain and difficult subscales (combined)
Mean change between EN3835 and placebo on the total score of the FFI pain and difficult subscales (combined) | Mean change from Baseline (Day 1) to Days15, 29, 43, and 57
  Mean change between EN3835 and placebo on the total score of the FFI pain and difficult subscales (combined)
Change in the proportion of EN3835-treated participants and those receiving only placebo reporting a 7-point scale Clinician Global Impression of Change Scale | Days 15, 29, 43, and 57
  Change in the proportion of EN3835-treated participants and those receiving only placebo reporting a 7-point scale Clinician Global Impression of Change Scale ranging from -3 ("Very Much Worse") to +3 ("Very Much Improvement")
Mean change between EN3835 and placebo in the nodular hardness of the treated nodules by durometer measurement | Baseline (Day 1) to Day 57
  Mean change between EN3835 and placebo in the nodular hardness of the treated nodules by durometer measurement
Mean change from Baseline in the nodular hardness of the treated nodules by durometer measurements with EN3835 vs placebo | Baseline (Day 1) to Days 15, 29, 43, 57
  Mean change from Baseline in the nodular hardness of the treated nodules by durometer measurements with EN3835 vs placebo
Safety of EN3835 as assessed by incidence, severity, and duration of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | Up to Day 57
  Safety of EN3835 as assessed by incidence, severity, and duration of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs)
Presence of anti-AUX-I and anti-AUX-II antibody titer levels in EN3835 treated participants | Day 1 and Day 57
  Presence of anti-AUX-I and anti-AUX-II antibody titer levels in EN3835 treated participants
Presence of neutralizing antibodies to AUX-I and AUX-II in EN3835 treated-participants | Day 1 and Day 57
  Presence of neutralizing antibodies to AUX-I and AUX-II in EN3835 treated-participants

CONTACTS AND LOCATIONS:
Overall Officials: Nina Green, Study Director — Endo Pharmaceuticals
Locations (43):
- United States (43):
  - Endo Clinical Trial Site #29, Mesa, Arizona
  - Endo Clinical Trial Site #42, Tucson, Arizona
  - Endo Clinical Trial Site #15, Bakersfield, California
  - Endo Clinical Trial Site #41, Encinitas, California
  - Endo Clinical Trial Site #9, Fresno, California
  - Endo Clinical Trial Site #27, La Mesa, California
  - Endo Clinical Trial Site #30, Los Angeles, California
  - Endo Clinical Trial Site #12, Tarzana, California
  - Endo Clinical Trial Site #36, Torrance, California
  - Endo Clinical Trial Site #22, Vista, California
  - Endo Clinical Trial Site #13, Whittier, California
  - Endo Clinical Trial Site #16, Atlantis, Florida
  - Endo Clinical Trial Site #43, Jacksonville, Florida
  - Endo Clinical Trial Site #40, Miami, Florida
  - Endo Clinical Trial Site #10, Pinellas Park, Florida
  - Endo Clinical Trial Site #3, South Miami, Florida
  - Endo Clinical Trial Site #14, Sweetwater, Florida
  - Endo Clinical Trial Site #38, Lawrenceville, Georgia
  - Endo Clinical Trial Site #31, Meridian, Idaho
  - Endo Clinical Trial Site #32, Decatur, Illinois
  - Endo Clinical Trial Site #19, O'Fallon, Illinois
  - Endo Clinical Trial Site #33, Springfield, Illinois
  - Endo Clinical Trial Site #23, Pasadena, Maryland
  - Endo Clinical Trial Site #28, Jefferson City, Missouri
  - Endo Clinical Trial Site #20, Las Vegas, Nevada
  - Endo Clinical Trial Site #34, Oklahoma City, Oklahoma
  - Endo Clinical Trial Site #4, York, Pennsylvania
  - Endo Clinical Trial Site #35, Arlington, Texas
  - Endo Clinical Trial Site #5, Bedford, Texas
  - Endo Clinical Trial Site #24, Cedar Park, Texas
  - Endo Clinical Trial Site #17, Dallas, Texas
  - Endo Clinical Trial Site #2, Dallas, Texas
  - Endo Clinical Trial Site #7, Fort Worth, Texas
  - Endo Clinical Trial Site #39, Georgetown, Texas
  - Endo Clinical Trial Site #25, Houston, Texas
  - Endo Clinical Trial Site #8, Houston, Texas
  - Endo Clinical Trial Site #1, McAllen, Texas
  - Endo Clinical Trial Site #21, San Antonio, Texas
  - Endo Clinical Trial Site #6, San Antonio, Texas
  - Endo Clinical Trial Site #18, Salt Lake City, Utah
  - Endo Clinical Trial Site #26, Lynchburg, Virginia
  - Endo Clinical Trial Site #37, Midlothian, Virginia
  - Endo Clinical Trial Site #11, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP